CLINICAL TRIAL: NCT03042858
Title: Natural History of Infants With Patent Processus Vaginalis
Acronym: HxPPV
Status: Recruiting | Type: Observational
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: Nationwide Children's Hospital (Other); C.S. Mott Children's Hospital (Other); University of Chicago (Other); James Whitcomb Riley Hospital for Children (Other); American Family Children's Hospital (Other); Children's Hospital and Health System Foundation, Wisconsin (Other); Norton Children's Hospital (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Shawn St. Peter, MD, Children's Mercy Hospital Kansas City
Other Study IDs: 16020156
Record Dates: First submitted 2017-02-01; First posted 2017-02-03 (Estimated); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Patent Processus Vaginalis; Inguinal Hernia
Keywords: PPV; patent processus vaginalis; inguinal hernia
MeSH Terms: conditions — Hernia, Inguinal | interventions — Predictive Value of Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (2):
- Infants with PPV: During laparoscopy for pyloric stenosis, the surgeon will turn the camera downward to answer the first question, whether the inguinal canal is patent or closed. If a PPV is present, the subject will be followed for up to 18 years of age.
  Interventions: Other: Infants with PPV
- Infants without PPV: During laparoscopy for pyloric stenosis, the surgeon will turn the camera downward to answer the first question, whether the inguinal canal is patent or closed. If there is no PPV, meaning they have normal anatomy, the patient demographic data will be recorded and this will terminate their participation.
  Interventions: Other: Infants without PPV

INTERVENTIONS:
Other: Infants with PPV — Data will be collected for up to 18 years to monitor for inguinal hernia.
  Groups: Infants with PPV
Other: Infants without PPV — Basic data will be collected regarding the surgery and the subject's study participation will be complete.
  Groups: Infants without PPV

SUMMARY:
This will be a multi-center prospective observational study of all patients who undergo laparoscopic pyloromyotomy. Subjects who have PPV will be followed up to just before their 18th birthday through annual phone calls or emails to determine the incidence and timing of subsequent inguinal hernia.

DETAILED DESCRIPTION:
Patients will be identified at the time the need for laparoscopic pyloromyotomy is determined by the consulting surgeon. After informed permission is obtained, demographic information will be collected on all subjects. Subjects who do not have PPV at the time of surgery will have no further data collected and their study participation will be complete. Subjects who have PPV will receive annual phone calls, emails, or other contact methods selected by the family, for up to before their 18th birthday or until they report having surgical inguinal hernia repair. Data will be recorded as noted on the master list and datasheet and entered into a REDCap database. All participating institutions will upload data into REDCap along with subject contact information so all follow up contact can be made by the coordinating center. All identifiable information in REDCap will be accessible by the coordinating center. Each enrolling center will have access to identifiers for their subjects only. Enrolling centers will be contacted and asked to update the contact information in REDCap if the coordinating center is not able to make contact with a subject. Subjects will also be given contact information for the coordinating center so they can provide updated information directly. Parents will be the main study contact for the duration of the study since no study interventions other than the phone call/email are required.

During laparoscopy for pyloric stenosis, the surgeon will turn the camera downward to answer the first question, whether the inguinal canal is patent or closed. Many surgeons routinely perform this maneuver; it takes no more than 10 seconds to perform and adds no risk to the operation. The study will include a quick estimate of width and depth of the PPV as outlined in the datasheet to characterize the size of the opening. The first characterization will be the presence of CO2 in the scrotum/labia upon insufflation, which clarifies that the PPV provides wide continuity from the abdomen to beyond the inguinal canal. The second characterization will be an estimate of the width of the opening in millimeters. The next step will be to note whether the bottom of the defect is seen. This is, by definition, no if the answer to the first question is yes and this no longer applies. Therefore the no answer to this question will identify those with an open tunnel but no external insufflation. Finally, if the bottom is seen then an estimate will be made in millimeters.

If there is no PPV, meaning the patient presents normal anatomy, the patient demographic data will be recorded and this will terminate their participation.

If a PPV is present, the investigators will conduct annual phone calls, or other contact method of the family's choice, to ask questions about whether the child has been diagnosed with hernia, underwent hernia repair or currently has symptoms consistent with a hernia (questionnaire attached). Subjects will be followed until hernia repair or as long as possible, up to their 18th birthday.

ELIGIBILITY:
Inclusion Criteria:

* All patients having laparoscopic surgery for pyloric stenosis. Subjects are anticipated to be less than four months of age at the time of enrollment.
* Enrollment inclusion dates: 08/2016 (upon IRB approval) to 7/31/2025

Exclusion Criteria:

* Patients who are anticipated to have a hostile abdomen for visualizing the inguinal rings (e.g. gastroschisis, necrotizing enterocolitis)
* Patients who have unilateral or bilateral undescended testes
* Patients undergoing open pyloromyotomy
* Patients who have a known hernia

Ages: 1 Day to 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants undergoing laparoscopic pyloromyotomy.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-01; Primary Completion 2035-12 (Estimated); Study Completion 2036-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of inguinal hernia | 18 years
  frequency of the development of symptomatic inguinal hernia in infants who are found to have an opening in their inguinal canal during laparoscopy for pyloric stenosis

SECONDARY OUTCOMES:
Time to development of inguinal hernia | 18 years
  Timeframe to develop a symptomatic inguinal hernia in infants who are found to have an opening in their inguinal canal during laparoscopy for pyloric stenosis.

CONTACTS AND LOCATIONS:
Overall Officials: Shawn D St. Peter, MD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
The data coordination site will have contact information for all subjects so that long-term follow-up can be done. Each contributing site will only have access to their own subjects' information.
Supporting Information: Study Protocol, Analytic Code
Time Frame: duration of study
Access Criteria: REDCap